CLINICAL TRIAL: NCT04649710
Title: A Double-Blind, Multicenter, Placebo-Controlled, Randomized, Parallel, Multiple-Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Pegbelfermin in Healthy Overweight and Obese Chinese and Korean Participants
Brief Title: A Study to Evaluate the Drug Levels and Safety of Pegbelfermin in Healthy Overweight and Obese Chinese and Korean Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MB130-063
Record Dates: First submitted 2020-11-25; First posted 2020-12-02 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Healthy Participants
Keywords: Chinese; Ethnicity; Korean; Obese; Overweight; Pegbelfermin
MeSH Terms: conditions — Obesity; Overweight | interventions — Pegbelfermin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort 1: Dose 1 or placebo (Experimental): Chinese participants
  Interventions: Biological: BMS-986036; Other: Placebo
- Cohort 2: Dose 2 or placebo (Experimental): Chinese participants
  Interventions: Biological: BMS-986036; Other: Placebo
- Cohort 3: Dose 1 or placebo (Experimental): Korean participants
  Interventions: Biological: BMS-986036; Other: Placebo
- Cohort 4: Dose 2 or placebo (Experimental): Korean participants
  Interventions: Biological: BMS-986036; Other: Placebo

INTERVENTIONS:
Biological: BMS-986036 — Specified dose on specified days
  Other Names: Pegbelfermin
Other: Placebo — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and drug level of Pegbelfermin in healthy overweight and obese Chinese and Korean participants.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obese, but otherwise healthy Chinese and Korean participants, as determined by no clinically significant deviations from normal in medical history, physical examination, electrocardiograms (ECGs), and clinical laboratory determinations
* Additional criterion for Chinese participants: must be first generation Chinese (born in China and not living outside of China for > 10 years, and both parents are ethnically Chinese)
* Additional criterion for Korean participants: must be first generation Korean (born in Korea and not living outside of Korea for > 10 years, and both parents are ethnically Korean)
* Must agree to follow specific methods of contraception, if applicable

Exclusion Criteria:

* BMI ≥ 40 kg/m^2
* Women who are pregnant or breastfeeding
* History of allergy to pegylated compounds or fibroblast growth factor 21-related compounds

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-21 (Estimated); Primary Completion 2021-09-21 (Estimated); Study Completion 2021-09-22 (Estimated)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of C-terminal intact BMS-986036 in Chinese and Korean participants | Up to 7 days after first dose and up to 7 days after last dose
Time of maximum observed plasma concentration (Tmax) of C-terminal intact BMS-986036 in Chinese and Korean participants | Up to 7 days after first dose and up to 7 days after last dose
Area under the concentration-time curve over 1 dosing interval (AUC (TAU)) of C-terminal intact BMS-986036 in Chinese and Korean participants | Up to 7 days after first dose and up to 7 days after last dose

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 45 days
Incidence of serious adverse events (SAEs) | Up to 70 days
Incidence of clinically significant changes in vital signs: Body temperature | Up to 64 days
Incidence of clinically significant changes in vital signs: Respiratory rate | Up to 64 days
Incidence of clinically significant changes in vital signs: Blood pressure | Up to 64 days
Incidence of clinically significant changes in vital signs: Heart rate | Up to 64 days
Incidence of clinically significant changes in physical examination findings | Up to 64 days
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: PR interval | Up to 64 days
  PR interval is the time from the onset of the P wave to the start of the QRS complex
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QRS | Up to 64 days
  QRS can be defined as the electrical impulse as it spreads through the ventricles, indicating ventricular depolarization
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QT interval | Up to 64 days
  The QT interval is the time from the start of the Q wave to the end of the T wave
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QTcF | Up to 64 days
  QTcF = Corrected QT interval using the Fridericia formula. QT interval is the time from the start of the Q wave to the end of the T wave
Incidence of clinically significant changes in clinical laboratory values: Hematology tests | Up to 64 days
Incidence of clinically significant changes in clinical laboratory values: Clinical chemistry tests | Up to 64 days
Incidence of clinically significant changes in clinical laboratory values: Urinalysis tests | Up to 64 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Local Institution, Changchun, Jilin, China
- Local Institution, Busan, South Korea

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm